CLINICAL TRIAL: NCT07395427
Title: Comparison of the Effects of Basic Body Awareness Therapy to Conventional Physiotherapy and Home Exercise Program in Individuals With Knee Osteoarthritis
Brief Title: Comparison of the Effects of Basic Body Awareness Therapy in Individuals With Knee Osteoarthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Emine Esra DİKMEN, Msc Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-FTR-EED-01
Record Dates: First submitted 2026-01-22; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; mind-body therapy; exercise; proprioception; physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised Control Clinical Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): BBAT plus home exercise programme
  Interventions: Other: BBAT plus home exercise programme
- Group B (Active Comparator): Conventional physiotherapy plus home exercise programme
  Interventions: Other: Conventional physiotherapy plus home exercise programme
- Group C (Active Comparator): Home exercise programme
  Interventions: Other: Home exercise programme

INTERVENTIONS:
Other: BBAT plus home exercise programme — The participants will undergo Basic Body Awareness Therapy (BBAT) for a total of 12 sessions, conducted as two non-consecutive sessions per week over a 6-week period. Each active exercise session will last between 30 and 45 minutes. The body awareness training will specifically focus on lower extremity exercises and will follow a progressive protocol. The program will commence with 5 exercises in the first week, adding one new exercise each week to reach a total of 10 BBAT exercises. Initially, repetitions will be set at 5; subsequently, each exercise will be adjusted to range between 5 and 10 repetitions. In addition to the supervised treatment, participants will be requested to perform home exercises at home at least 3 days a week as 2 sets for a duration of 8 weeks, and an exercise diary will be provided. Prior to the treatment, the importance and content of the exercises will be thoroughly explained.
  Arms: Group A
Other: Conventional physiotherapy plus home exercise programme — Before each treatment session, a hot pack (thermotherapy) will be applied to the knee, calf, and thigh muscles for 20 minutes, followed by therapeutic ultrasound administered to the periarticular knee region for 10 minutes in pulsed mode, with a frequency of 1.0 MHz, an intensity of <1 W/cm², and a total dose of <150 J/cm². Exercises and recommendations identical to those prescribed for the home exercise group will be explained to the patients, and they will be instructed to perform these exercises in addition to the treatment, for 8 weeks, at least 3 days per week, in 2 sets per session. An exercise diary will be provided to monitor adherence. Prior to treatment, participants will be informed about the importance and content of the exercise program.
  Other Names: traditional physiotherapy; classic physiotherapy
  Arms: Group B
Other: Home exercise programme — Based on the guidelines published by the American College of Sports Medicine (ACSM), Osteoarthritis Research Society International (OARSI), American Academy of Orthopaedic Surgeons (AAOS), European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO), and the European Alliance of Associations for Rheumatology (EULAR), participants will be prescribed a total of 12 home-based exercises to be performed over 8 weeks, at least 3 days per week, in 2 sets per session, with the number of repetitions progressively increased .
  These exercises and recommendations will be categorized under the subheadings of aerobic exercise, muscle strengthening, flexibility, neuromotor performance, and patient education. To enhance exercise adherence and facilitate follow-up, participants will be provided with an exercise diary. The diary will include a 3-month calendar schedule, illustrations of the exercises, and coded numerical markers correspo
  Other Names: home-based exercise programme
  Arms: Group C

SUMMARY:
Osteoarthritis (OA) is a chronic, degenerative joint disease associated with aging and is recognized by the World Health Organization as a primary health condition. It is one of the leading causes of chronic disability worldwide. Structural changes occurring at the bone and joint margins in OA lead to a variety of symptoms and clinical findings associated with the deterioration of articular cartilage integrity.

Clinical guidelines recommend a combination of exercise therapy tailored to individual needs, weight loss, and patient education prior to considering arthroplasty. However, achieving satisfactory long-term outcomes remains challenging, as patients are often unmotivated to adhere to training programs involving functional strength and mobility exercises unless they are supervised by a physiotherapist. Basic Body Awareness Therapy (BBAT) may serve as an alternative exercise method with a higher potential for sustained effects.

BBAT is a movement-based therapy applied to daily life activities, focusing on body alignment and movement quality. Through the learning process of BBAT-by doing, reflecting, and transferring body awareness into everyday movements-it is hypothesized that patients gain self-efficacy and skills essential for maintaining independent and continuous exercise. BBAT is a body-mind therapeutic approach that emphasizes awareness of body sensations and movement patterns, aiming to restructure body awareness and motor control through individual experience. Increased attention to movement and bodily experiences enhances awareness of both physical and mental aspects.

Through specific exercises, BBAT helps to reveal and improve the interaction and synergy between body and mind, thereby promoting postural stability, movement fluidity, and awareness of bodily reactions and internal resources. By encouraging reduced energy expenditure during daily activities and improving movement quality through self-exploration and experiential learning, BBAT contributes to improvements in postural imbalance, muscle tension, and bodily dysfunction. BBAT movements are simple, comfortable, balanced, and based on repeated experiential learning. Exercises are performed in various positions, including lying, sitting, standing, and walking. Physiotherapists guide patients using both physical and verbal cues to facilitate improved postural control, balance, and breathing during movement.

Central sensitization may lead individuals with osteoarthritis to perceive normal bodily functions as painful, resulting in compensatory and dysfunctional movement strategies. It has been reported that mindfulness-based and body-mind therapies can reduce pain and symptoms while improving physical function in clinical management. Moreover, as emphasized in the recommendations of the Osteoarthritis Research Society International (OARSI), active patient involvement in health management is a core component of body-mind therapies such as BBAT.

Despite these potential benefits, there is a limited number of studies investigating the effects of BBAT in individuals with osteoarthritis. Given that BBAT requires no equipment, can be practiced in any setting, promotes social engagement through group-based sessions, enhances relaxation and mind-body awareness, and reduces stress and anxiety, it may represent a favorable alternative exercise model. Additionally, BBAT may improve exercise adherence and contribute to reducing healthcare burden and associated costs. Comparing the effects of different therapeutic programs across multiple outcome parameters may help identify the most effective interventions for individuals with osteoarthritis, thereby improving clinical outcomes.

In this context, the present study aims to compare the effects of Basic Body Awareness Therapy, applied in addition to conventional physiotherapy and a home exercise program, on pain, muscle strength, range of motion, balance, active joint position sense, functional outcomes, pressure pain threshold, kinesiophobia, and quality of life in individuals with knee osteoarthritis.

DETAILED DESCRIPTION:
This study is designed as a three-arm randomized controlled clinical trial to evaluate the effectiveness of Basic Body Awareness Therapy (BBAT) compared with conventional physiotherapy and a home exercise program in individuals with knee osteoarthritis. Eligible participants will be randomly allocated to one of three intervention groups: (1) BBAT plus home exercise, (2) conventional physiotherapy plus home exercise, or (3) home exercise only.

The intervention period will last six weeks, with a total program duration of eight weeks. BBAT and conventional physiotherapy interventions will be delivered twice weekly by licensed physiotherapists according to standardized treatment protocols. BBAT sessions will be conducted in group settings and will focus on body awareness, posture, breathing, and controlled movement patterns. Participants in all groups will follow the same structured home exercise program.

Outcome assessments will be conducted at baseline and after completion of the intervention period. Primary and secondary outcomes will include pain intensity, proprioception, functional status, balance, physical performance, muscle strength, joint range of motion, edema, fatigue, kinesiophobia, and quality of life. These outcomes will be evaluated using validated clinical assessment methods and patient-reported outcome measures.

The primary objective of this study is to compare the effects of BBAT, conventional physiotherapy, and home exercise on clinical and functional outcomes in individuals with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Grade 2-3 knee osteoarthritis based on the Kellgren-Lawrence radiographic grading system.
* Aged between 40 and 74 years.
* Meeting the clinical classification criteria of the American College of Rheumatology (ACR).

Exclusion Criteria:

* Current or previous history of malignancy.
* Pregnancy or lactation.
* History of prior surgical intervention involving the knee or hip joints.
* Presence of neurological disorders impacting the innervation of the hip or knee musculature.
* Presence of concomitant inflammatory or infectious pathologies localized to the hip or knee joints.
* Having undergone physical therapy or rehabilitation interventions within the preceding 6 months.
* Administration of intra-articular injections (PRP, GRP, stem cell or corticosteroids) within the last 6 months.
* Severe cognitive impairment or diagnosis of dementia.
* Participation in regular physical exercise or sports activities for a minimum of 3 days per week.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength / Hand-held dinamometer - Lafayette Instrument®, Lafayette, IN | 8 weeks
  Lower extremity muscle strength will be evaluated using a hand-held dynamometer (Lafayette Instrument®, Lafayette, IN) via maximal voluntary isometric contraction (the "make" test) and recorded in kilograms/Newtons. The assessment will include the muscle strength of hip flexion, extension, abduction, adduction, external and internal rotation; knee flexion and extension; and ankle plantar/dorsi flexion. Participants will be given the command: 'Hold as strongly as possible without moving your leg.' For each movement, three measurements will be performed (5-second contraction, 30-second rest), and the average values of these measurements will be calculated.
Balance - Fullerton Advanced Balance Scale (FAB-T) | 8 weeks
  The scale evaluates both static and dynamic balance under altered sensory conditions (soft surface, firm surface, decreased or increased support base, and verbal commands). It is specifically designed to measure balance in high-functioning, active older adults. The scale consists of 10 items, each scored between 0 and 4. A total score of 25 or below indicates a high risk of falling.
Pain Severity - The Numerical Rating Scale (NRS) | 8 weeks
  Pain severity over the past 24 hours (at its worst, at its best, and at rest) will be assessed via the Numeric Rating Scale (NRS) on a scale of 0 to 10, where 0 represents 'no pain' and 10 represents 'the worst imaginable pain.
Active Joint Position Sense (AJPS) | 8 weeks
  AJPS will be evaluated via photo-analysis using MATLAB and an iPhone 13 (50 cm distance, tripod, laser alignment). Anatomical markers (2x2 cm kinesio-tape) will be placed on the greater trochanter, lateral knee joint line, superior patella, fibular neck, and lateral malleolus. Participants in the supine position, with hips neutral and eyes masked, will actively reproduce target knee flexion angles (40°, 60°, 90°). Reference and reproduced positions will be photographed; the angular difference will be recorded as the error angle. After practice trials, measurements will be captured during a 4-second static phase. Three trials per angle will be performed in randomized order with 10-second intervals, and averages will be calculated. To prevent fatigue and angular memory bias, 1-minute rest periods will be provided. All measurements will be standardized by an experienced physiotherapist.
Knee Function (KOOS) | 8 weeks
  Knee Injury and Osteoarthritis Outcome Score (KOOS): Developed to assess knee injury and OA symptoms. It includes 42 items in 5 subscales: Pain, Symptoms, ADL, Sport/Rec, and QoL. Items are scored on a 0-4 Likert scale based on the past week. Each subscale is normalized to a 0-100 range.
Physical Mobility - TUG Test | 8 weeks
  Timed Up and Go (TUG) Test: TUG assesses independent mobility and functional ability. Participants rise from a chair, walk 3 meters at a safe pace, turn, walk back, and sit down. The duration is recorded in seconds.
  Results are interpreted as follows: ≤10 seconds indicates good balance and gait speed; 10-20 seconds indicates independence in outdoor mobility without aids; ≥20 seconds signifies impaired mobility, poor balance, and increased fall risk. The test provides a reliable measure of dynamic balance and functional performance in clinical populations. All procedures will be timed using a digital stopwatch and recorded.
Pressure Pain Threshold (PPT)/ (JTECH Medical-Algometer Commander, USA) | 8 weeks
  Measurements will be performed while the participant is in the supine and prone positions using a pressure algometer. In the supine position, measurements will be taken from the distal 1/3 of the iliopsoas muscle, the proximal and distal (suprapatellar) portions of the rectus femoris muscle, the infrapatellar tendon, the medial and lateral fat pads, the distal 1/3 of the iliotibial band, the adductor tendons, and the medial retinaculum. In the prone position, measurements will be obtained from the sacroiliac joint, the muscle bellies of the gluteus medius and piriformis, the proximal 1/3 of the medial and lateral heads of the gastrocnemius, and the popliteus muscle belly. The probe of the algometer will be applied perpendicularly to the designated area, and the pressure will be increased gradually at a rate of 1 kg/s. The value at which the mechanical stimulus first transitions into a sensation of pain will be recorded. Three measurements will be taken at 30-second intervals.
The Pain Catastrophizing Scale (PCS) | 8 weeks
  Pain Catastrophizing Scale (PCS): A 13-item self-report tool used to measure exaggerated negative thoughts about actual or anticipated pain. It assesses three dimensions: Rumination (items 8-11), Magnification (items 6, 7, 13), and Helplessness (items 1-5, 12). Rumination reflects preoccupation with pain, helplessness denotes an inability to cope, and magnification represents an intensified perception of pain threat.
  Each item is rated on a 5-point Likert scale (0=not at all, 4=all the time). Total scores range from 0 to 52, where higher scores indicate greater catastrophizing. A total score of ≥30 is identified as the clinical cutoff point for significant pain catastrophizing. This scale is vital for evaluating the psychological impact of pain and its influence on recovery and movement-related fear in clinical research and rehabilitation settings.
Knee Function (LYSHOLM) | 8 weeks
  Lysholm Knee Scoring Scale: Revised in 1985, it assesses 8 domains: limp, support, locking, instability, pain, swelling, stair climbing, and squatting. Total score (0-100) is categorized as Excellent (95-100), Good (84-94), Fair (65-83), or Poor (0-64).
Knee Function (WOMAC) | 8 weeks
  Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC): A valid index for OA, recommended by OMERACT. It comprises 24 items across 3 sections: Pain (max 20), Stiffness (max 8), and Physical Function (max 68). Higher scores indicate increased pain, stiffness, and functional impairment. All scales will be administered by a physiotherapist to evaluate functional status and quality of life.

SECONDARY OUTCOMES:
Quality of Life / (World Health Organization Quality of Life Scale - Brief Form (WHOQOL-BREF) | 8 weeks
  WHOQOL-BREF: A 26-item cross-cultural tool assessing four domains: physical, psychological, social relationships, and environment. It includes two general items on perceived health and quality of life. Domains are scored from 0 to 100, where higher scores indicate better well-being.
Kinesiophobia - Tampa Scale for Kinesiophobia (TSK) | 8 weeks
  The scale consists of 17 items designed to measure the fear of movement and (re)injury. It utilizes a 4-point Likert scale (1: Strongly disagree, 2: Disagree, 3: Agree, 4: Strongly agree). Items 4, 8, 12, and 16 are reverse-scored. Total scores range from 17 to 68, where higher scores indicate a greater degree of kinesiophobia (fear of movement).
Aerobic and Physical Performance (Stair Climb Test) | 8 weeks
  A staircase consisting of 9 steps (16-20 cm height) with handrails will be used. Participants will be instructed to ascend and descend as quickly and safely as possible. The total completion time will be recorded in seconds. This test provides data on lower extremity muscle strength and balance.
Edema Assesment (Tape Measure) | 8 weeks
  Edema assessment will be performed using the circumference measurement technique with a foldable, non-elastic, 7-mm wide tape measure. To ensure the measurement is unaffected by tension, the starting end of the tape will be held in the left hand while the other end is wrapped around the limb with the right hand, and the value aligning with the starting point will be recorded. Furthermore, during measurement, the starting point and the corresponding value will be aligned side-by-side rather than overlapping. Participants will wear shorts to facilitate the identification of anatomical landmarks. Since the patella is the reference point for the thigh, measurements will be taken from the mid-patella, as well as 5 and 10 cm superiorly and inferiorly from both legs. To minimize potential errors arising from incorrect positioning or varying tension, all measurements will be performed by the same researcher to ensure inter-rater reliability.
Range of Motion (ROM) - (Universal Goniometer) | 8 weeks
  Goniometric Assessment: AROM and PROM of the hip and knee will be measured using standardized protocols. Hip flexion (supine, knee flexed) and extension (prone, knee extended) use the greater trochanter as the fulcrum. Abduction and adduction (supine) align the stationary arm with the ASIS line. Internal and external rotation are assessed in the sitting position with the fulcrum at the tibial tuberosity and the stationary arm perpendicular to the floor. Knee flexion is measured in the prone position with the fulcrum at the lateral femoral condyle. Precautions include maintaining pelvic stability and preventing compensatory movements such as lumbar lordosis or pelvic elevation. All measurements start from a 0° neutral position. This comprehensive 2026 clinical evaluation ensures precise documentation of joint mobility, essential for monitoring rehabilitation progress and functional recovery in musculoskeletal physical therapy.
Fatique / Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | 8 weeks
  The FACIT-F is a 13-item self-report scale designed to evaluate fatigue and its impact on daily activities and functions. Originally developed to assess the relationship between anemia and fatigue in cancer patients, its validity and reliability have since been established across more than 70 published studies involving over 20,000 participants. Since 1995, it has been proven effective for various conditions, including Multiple Sclerosis, Rheumatoid Arthritis, Psoriasis, Parkinson's disease, and Paroxysmal Nocturnal Hemoglobinuria. The scale measures the level of fatigue experienced during the past 7 days. Each item is rated on a 5-point Likert scale (0: Not at all, 4: Very much). Total scores range from 0 to 52, where higher scores indicate lower levels of fatigue. Items 1, 2, 3, 4, 5, 6, 9, 10, 11, 12, and 13 are reverse-scored, while items 7 and 8 are scored directly. It is a cross-culturally validated tool approved for use in adults with chronic illnesses.
World Health Organization Quality of Life - Older Adults Module (WHOQOL-OLD) | 8 weeks
  WHOQOL-OLD: A 24-item module specifically for older adults, consisting of six facets: Sensory Abilities, Autonomy, Past/Present/Future Activities, Social Participation, Death and Dying, and Intimacy. Items use a 5-point Likert scale, with facet scores ranging from 4 to 20. It evaluates the impact of aging on independence, social engagement, and mortality concerns. Increased total scores represent improved quality of life. Both scales provide a multidimensional profile of the participant's subjective well-being and are validated in Turkish. These instruments are essential for evaluating the holistic outcomes of geriatric rehabilitation and 2026 clinical standards in elderly care.
Aerobic and Physical Performance (6-Minute Walk Test (6MWT)) | 8 weeks
  The 6MWT is a submaximal exercise test used to evaluate aerobic capacity and endurance. The distance covered over 6 minutes is recorded. A 30-meter unobstructed corridor, cones, and a stopwatch are required. Participants may rest if needed, but the timer continues. Dyspnea intensity will be assessed using the Modified Borg Scale before and after the test. The Modified Borg Scale is a 0-10 rating scale (0: None, 10: Maximum) used to measure perceived exertion and dyspnea severity. It is highly reliable for determining exercise intensity and monitoring subjective fatigue pre- and post-session.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University/Faculty of Physical Therapy and Rehabilitation/ Orthopedic Rehabilitation Unit, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual patient-level data are not publicly available due to privacy and confidentiality considerations. Individual participant data were not shared because they contain confidential and potentially identifiable information, and data sharing was not covered by the informed consent obtained from participants. Therefore, access to these data is restricted in accordance with ethical standards and data protection regulations.

REFERENCES:
- [Background] Singh H, Arya S, Talapatra P, Lather K, Mathur R, Singhania A, Chaudhary V. Assessment of fatigue in rheumatoid arthritis (by Functional Assessment of Chronic Illness Therapy-Fatigue score) and its relation to disease activity and anemia. J Clin Rheumatol. 2014 Mar;20(2):87-90. doi: 10.1097/RHU.0000000000000073. PMID 24561411
- [Background] Eser S, Saatli G, Eser E, Baydur H, Fidaner C. [The reliability and validity of the Turkish Version of the World Health Organization Quality of Life Instrument-Older Adults Module (WHOQOL-Old)]. Turk Psikiyatri Derg. 2010 Spring;21(1):37-48. Turkish. PMID 20204903
- [Background] Power M, Quinn K, Schmidt S; WHOQOL-OLD Group. Development of the WHOQOL-old module. Qual Life Res. 2005 Dec;14(10):2197-214. doi: 10.1007/s11136-005-7380-9. PMID 16328900
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Vlaeyen JW, Kole-Snijders AM, Rotteveel AM, Ruesink R, Heuts PH. The role of fear of movement/(re)injury in pain disability. J Occup Rehabil. 1995 Dec;5(4):235-52. doi: 10.1007/BF02109988. PMID 24234727
- [Background] Tuzun EH, Eker L, Aytar A, Daskapan A, Bayramoglu M. Acceptability, reliability, validity and responsiveness of the Turkish version of WOMAC osteoarthritis index. Osteoarthritis Cartilage. 2005 Jan;13(1):28-33. doi: 10.1016/j.joca.2004.10.010. PMID 15639634
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Celik D, Coskunsu D, Kilicoglu O. Translation and cultural adaptation of the Turkish Lysholm knee scale: ease of use, validity, and reliability. Clin Orthop Relat Res. 2013 Aug;471(8):2602-10. doi: 10.1007/s11999-013-3046-z. Epub 2013 May 11. PMID 23666590
- [Background] Lysholm J, Gillquist J. Evaluation of knee ligament surgery results with special emphasis on use of a scoring scale. Am J Sports Med. 1982 May-Jun;10(3):150-4. doi: 10.1177/036354658201000306. PMID 6896798
- [Background] Gul ED, Yilmaz O, Bodur H. Reliability and validity of the Turkish version of the knee injury and osteoarthritis outcome score-physical function short-form (KOOS-PS). J Back Musculoskelet Rehabil. 2013;26(4):461-6. doi: 10.3233/BMR-130406. PMID 23948834
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Darnall BD, Sturgeon JA, Cook KF, Taub CJ, Roy A, Burns JW, Sullivan M, Mackey SC. Development and Validation of a Daily Pain Catastrophizing Scale. J Pain. 2017 Sep;18(9):1139-1149. doi: 10.1016/j.jpain.2017.05.003. Epub 2017 May 19. PMID 28528981
- [Background] Arden NK, Perry TA, Bannuru RR, Bruyere O, Cooper C, Haugen IK, Hochberg MC, McAlindon TE, Mobasheri A, Reginster JY. Non-surgical management of knee osteoarthritis: comparison of ESCEO and OARSI 2019 guidelines. Nat Rev Rheumatol. 2021 Jan;17(1):59-66. doi: 10.1038/s41584-020-00523-9. Epub 2020 Oct 28. PMID 33116279
- [Background] Skou ST, Roos EM. Physical therapy for patients with knee and hip osteoarthritis: supervised, active treatment is current best practice. Clin Exp Rheumatol. 2019 Sep-Oct;37 Suppl 120(5):112-117. Epub 2019 Oct 15. PMID 31621559
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Care Res (Hoboken). 2020 Feb;72(2):149-162. doi: 10.1002/acr.24131. Epub 2020 Jan 6. PMID 31908149
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Fernandes L, Hagen KB, Bijlsma JW, Andreassen O, Christensen P, Conaghan PG, Doherty M, Geenen R, Hammond A, Kjeken I, Lohmander LS, Lund H, Mallen CD, Nava T, Oliver S, Pavelka K, Pitsillidou I, da Silva JA, de la Torre J, Zanoli G, Vliet Vlieland TP; European League Against Rheumatism (EULAR). EULAR recommendations for the non-pharmacological core management of hip and knee osteoarthritis. Ann Rheum Dis. 2013 Jul;72(7):1125-35. doi: 10.1136/annrheumdis-2012-202745. Epub 2013 Apr 17. PMID 23595142
- [Background] Sale JE, Gignac M, Hawker G. The relationship between disease symptoms, life events, coping and treatment, and depression among older adults with osteoarthritis. J Rheumatol. 2008 Feb;35(2):335-42. Epub 2008 Jan 15. PMID 18203312
- [Background] Lluch E, Nijs J, Courtney CA, Rebbeck T, Wylde V, Baert I, Wideman TH, Howells N, Skou ST. Clinical descriptors for the recognition of central sensitization pain in patients with knee osteoarthritis. Disabil Rehabil. 2018 Nov;40(23):2836-2845. doi: 10.1080/09638288.2017.1358770. Epub 2017 Aug 2. PMID 28768437
- [Background] Skjaerven LH, Mattsson M, Catalan-Matamoros D, Parker A, Gard G, Gyllensten AL. Consensus on core phenomena and statements describing Basic Body Awareness Therapy within the movement awareness domain in physiotherapy. Physiother Theory Pract. 2019 Jan;35(1):80-93. doi: 10.1080/09593985.2018.1434578. Epub 2018 Feb 26. PMID 29482403
- See also: American Academy of Orthopaedic Surgeons Management of Osteoarthritis of the Knee (Non-Arthroplasty) Evidence-Based Clinical Practice Guideline — https://www.aaos.org/oak3cpg

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2026-01-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT07395427/Prot_SAP_ICF_000.pdf